CLINICAL TRIAL: NCT02878135
Title: the Effect of Slow Versus Fast Application of Vulsellum on Pain Perception During Intrauterine Device Insertion
Brief Title: Fast Versus Slow Application of Vulsellum During Intrauterine Device Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SLVOL
Record Dates: First submitted 2016-08-22; First posted 2016-08-25 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Improving Quality of Life

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- fast vulsellum (Experimental): rapid ratchet of the vulsellum
  Interventions: Procedure: fast application
- slow vulsellum (Active Comparator): Placement of the tenaculum over 7-10 seconds and not allowing the vulsellum to ratchet audibly.
  Interventions: Procedure: slow application

INTERVENTIONS:
Procedure: fast application
  Arms: fast vulsellum
Procedure: slow application
  Arms: slow vulsellum

SUMMARY:
intrauterine device insertion requires use a vulsellum to stabilize the cervix. Patient's often complain that its placement is one of the most uncomfortable parts of this procedure

ELIGIBILITY:
Inclusion Criteria:

* Women not taken analgesics or anxiolytics in the 24 hours prior insertion
* Women not taken misoprostol prior to intrauterine device insertion
* Women who will accept to participate in the study

Exclusion Criteria:

Any contraindication to intrauterine device placement

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
mean Pain score with vulsellum placement | 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abbas, MD, Principal Investigator — Assiut University
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes